CLINICAL TRIAL: NCT04979351
Title: The Effect of Post Colonoscopy Abdominal Massage on Abdominal Pain, Distension, Discomfort and Patient Satisfaction: a Randomized Controlled Study Protocol
Brief Title: The Effect of Post Colonoscopy Abdominal Massage on Abdominal Pain, Distension, Discomfort and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Dilek Ozturk, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CemilTascıogluERHO
Record Dates: First submitted 2021-07-10; First posted 2021-07-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Colonoscopy; abdominal massage; abdominal pain; abdominal distension; abdominal discomfort; patient satisfaction
MeSH Terms: conditions — Abdominal Pain; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abdominal Massage Group (Experimental): Abdominal massage for 15 minutes twice a day application.
  Interventions: Other: Abdominal Massage
- Placebo Group (No Intervention): Abdominal massage was not applied.

INTERVENTIONS:
Other: Abdominal Massage — Abdominal massage will be applied twice a day.
  Arms: Abdominal Massage Group

SUMMARY:
Background: Abdominal pain, distension, and discomfort are the most frequently seen side effects after colonoscopy. These side effects can cause physical and mental results and increased workloads and care costs. Additionally, the satisfaction of the patients with the colonoscopy process may affect their willingness to undergo repeated colonoscopies in the future which may be required for the surveillance of colon malignity. Currently, there are no studies evaluating the effects of abdominal massage on post colonoscopy these abdominal symptoms. The aim of this study was to evaluate the effect of post colonoscopy abdominal massage on abdominal pain, distension, discomfort, and patient satisfaction.

Methods: This study was designed as a prospective randomized controlled study. Participants meeting inclusion criteria will be assigned to intervention and control groups using a random number generator. Participants assigned to the intervention group will receive abdominal massages twice a day after colonoscopy, and participants assigned to the control group will receive only "routine care". The abdominal pain, distension, discomfort, and satisfaction levels of the patients will be evaluated using the Visual Analogue Scale.

Conclusions: New approaches are needed to improve the physiological and psychological health levels of patients after colonoscopy and help them return to their daily life activities and social lives faster. The trial will provide valuable evidence to inform clinical application and help evaluate the effects of the use of the relevant intervention.

DETAILED DESCRIPTION:
Abdominal pain, bloating, and discomfort are the most frequently problems experienced by patients undergoing colonoscopy. These problems are thought to be caused by several factors such as the duration of the process, the technical difficulty level of the process, distension caused by air insufflation, and the expertise level of the endoscopist. These problems are experienced by approximately a third of patients undergoing colonoscopy, and may last from a few hours to a few days. In a recent study, 44% of patients were found to experience such minor side effects 24 hours after colonoscopy, and 23% were found to experience them after a 30 day follow up. Although these problems are dubbed minor side effects, they may cause serious results for patients with regard to physical comfort and mental stress and may necessitate patients to be monitored post colonoscopy and followed up closely. This may lead to an increase in costs by increasing the length of hospital stay and nursing care requirements. Additionally, the satisfaction of the patients with the colonoscopy process may affect their willingness to undergo repeated colonoscopies in the future which may be required for the surveillance of colon malignity. For these reasons, decreasing post colonoscopy abdominal pain, distension, and discomfort and increasing patient satisfaction may increase the acceptance of future colonoscopy screening for colorectal cancers.

Studies focused on decreasing abdominal symptoms after colonoscopy and increasing patient comfort and satisfaction have yielded varying results. For example, while some studies have reported that rectal tube application after colonoscopy reduces pain and increases patient comfort and satisfaction, in another study, it was determined that rectal tube application post colonoscopy had no effect on abdominal distension, pain, discomfort, and patient satisfaction after the process and 24 hours later. In another study, rectal aspiration applied right after colonoscopy was found to be more effective in decreasing abdominal symptoms compared to the application of rectal tubes after colonoscopy. In another study where total colonic decompression through repeating cecal intubation after colonoscopy was applied, the method was found to decrease the distension complaints of patients in the early post colonoscopy period from 59% to 25%. However, in this study, no significant difference between the groups that did and did not receive decompression with regard to abdominal pain and distension could be found 24 to 48 hours after the procedure. In yet another study, no significant difference with regard to pain intensity could be found between the aspiration of air in the curves of the colon without repeated intubation while the colonoscope was being taken out and rectal aspiration.

Abdominal massaging has been shown to help improve symptoms in patients with severe constipation. In the literature, it has been reported that abdominal massage relaxes the abdominal muscles and stimulates the excretory activity by supporting the intestine, decrease discomfort and pain in individuals with abdominal pain related to cramps or flatulence, and increase the quality of life. Moreover, it is a non-invasive and safe non-pharmacological method. It has no known side effects and does not require any cost.

In this study, it was assumed post-colonoscopy abdominal massage can improve their abdominal symptoms. However, to date, there is no study evaluating the effects of abdominal massage on abdominal symptoms after colonoscopy. Therefore, a prospective study was designed to evaluate the aspect of post-colonoscopy abdominal massage that concerns endoscopy nurses, namely its effect on abdominal pain, bloating, discomfort and patient satisfaction.

Aim

The aim of this study was to evaluate the effect of post colonoscopy abdominal massage on abdominal pain, distension, discomfort, and patient satisfaction.

Null hypothesis

There will be no significant difference between patients receiving abdominal massage post colonoscopy and those not receiving such an intervention with regard to abdominal pain, distension, discomfort, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* being of 18 years of age and above
* owning a cell phone
* having a body mass index below 30
* being conscious and having location
* people, and time orientation
* having no communication barriers
* being able to communicate in Turkish
* giving written informed consent to participate in the study

Exclusion Criteria:

* were receiving sedation
* having previously received intestine resection or other intestinal surgery
* having an uncontrolled psychopathological illness
* receiving colonoscopy for treatment
* having active lower gastrointestinal system bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | The end of the second day.
  Abdominal pain will be evaluated with the Visual Analog Scale Zero = minimum value Ten = maximum value

SECONDARY OUTCOMES:
Abdominal distension | The end of the second day.
  Abdominal distension will be evaluated with the Visual Analog Scale Zero = minimum value Ten = maximum value

OTHER OUTCOMES:
Comfort | The end of the second day.
  Abdominal comfort will be evaluated with the Visual Analog Scale Zero = minimum value Ten = maximum value
High Satisfaction | The end of the second day.
  Patient satisfaction will be evaluated with the Visual Analog Scale Zero = minimum value Ten = maximum value

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK ÖZTÜRK, MSc, Principal Investigator — specify Unaffiliated; Aysel GÜRKAN, PhD, Study Director — specify Unaffiliated
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study results will be shared.
Supporting Information: Study Protocol
Time Frame: No time limit
Access Criteria: No Access Criteria

REFERENCES:
- [Background] Steffenssen MW, Al-Najami I, Zimmermann-Nielsen E, Baatrup G. Patient-reported complications related to colonoscopy: a prospective feasibility study of an email-based survey. Acta Oncol. 2019;58(sup1):S65-S70. doi: 10.1080/0284186X.2018.1535188. Epub 2018 Dec 7. PMID 30523730
- [Background] Sumanac K, Zealley I, Fox BM, Rawlinson J, Salena B, Marshall JK, Stevenson GW, Hunt RH. Minimizing postcolonoscopy abdominal pain by using CO(2) insufflation: a prospective, randomized, double blind, controlled trial evaluating a new commercially available CO(2) delivery system. Gastrointest Endosc. 2002 Aug;56(2):190-4. doi: 10.1016/s0016-5107(02)70176-4. PMID 12145595
- [Background] Erstad DJ, Krowsoski LS, Kaafarani HM. Abdominal Pain After Colonoscopy. Gastroenterology. 2017 Feb;152(3):486-487. doi: 10.1053/j.gastro.2016.08.060. Epub 2017 Jan 3. No abstract available. PMID 28056353
- [Background] Yi CH, Liu TT, Lei WY, Hung JS, Chen CL. Influence of Rectal Decompression on Abdominal Symptoms and Anorectal Physiology following Colonoscopy in Healthy Adults. Gastroenterol Res Pract. 2016;2016:4101248. doi: 10.1155/2016/4101248. Epub 2016 Aug 29. PMID 27651788
- [Background] Liu TT, Yi CH, Lei WY, Yu HC, Hung JS, Chen CL. Comparison of rectal suction versus rectal tube insertion for reducing abdominal symptoms immediately after unsedated colonoscopy. Endosc Int Open. 2016 Jun;4(6):E725-9. doi: 10.1055/s-0034-1392223. Epub 2015 Dec 15. PMID 27336061
- [Background] Devitt J, Shellman L, Gardner K, Nichols LW. Using positioning after a colonoscopy for patient comfort management. Gastroenterol Nurs. 2011 Mar-Apr;34(2):93-100. doi: 10.1097/SGA.0b013e31820f9ac3. PMID 21455041
- [Background] Kim SY, Kim HS, Park HJ. Adverse events related to colonoscopy: Global trends and future challenges. World J Gastroenterol. 2019 Jan 14;25(2):190-204. doi: 10.3748/wjg.v25.i2.190. PMID 30670909
- [Background] Lynch I, Hayes A, Buffum MD, Conners EE. Insufflation using carbon dioxide versus room air during colonoscopy: comparison of patient comfort, recovery time, and nursing resources. Gastroenterol Nurs. 2015 May-Jun;38(3):211-7. doi: 10.1097/SGA.0000000000000109. PMID 25946475
- [Background] Steinberg EN, Howden CW. Randomized controlled trial of rectal tube placement for the management of abdominal distension following colonoscopy. Gastrointest Endosc. 1997 Nov;46(5):444-6. doi: 10.1016/s0016-5107(97)70038-5. PMID 9402119
- [Background] Hilzenrat N, Fich A, Odes HS, Krugliak P, Eidelman L, Gaspar N, Weisberg G, Rosenthal A, Delgado JL, Ginat R, Sperber AD. Does insertion of a rectal tube after colonoscopy reduce patient discomfort and improve satisfaction? Gastrointest Endosc. 2003 Jan;57(1):54-7. doi: 10.1067/mge.2003.47. PMID 12518131
- [Background] Lee JG, Vigil H, Leung JW. A randomized controlled trial of total colonic decompression after colonoscopy to improve patient comfort. Am J Gastroenterol. 2001 Jan;96(1):95-100. doi: 10.1111/j.1572-0241.2001.03458.x. PMID 11197295
- [Background] Lamas K, Lindholm L, Stenlund H, Engstrom B, Jacobsson C. Effects of abdominal massage in management of constipation--a randomized controlled trial. Int J Nurs Stud. 2009 Jun;46(6):759-67. doi: 10.1016/j.ijnurstu.2009.01.007. Epub 2009 Feb 12. PMID 19217105
- [Background] Liu Z, Sakakibara R, Odaka T, Uchiyama T, Yamamoto T, Ito T, Hattori T. Mechanism of abdominal massage for difficult defecation in a patient with myelopathy (HAM/TSP). J Neurol. 2005 Oct;252(10):1280-2. doi: 10.1007/s00415-005-0825-9. Epub 2005 May 20. No abstract available. PMID 15895308
- [Background] Sinclair M. The use of abdominal massage to treat chronic constipation. J Bodyw Mov Ther. 2011 Oct;15(4):436-45. doi: 10.1016/j.jbmt.2010.07.007. Epub 2010 Aug 25. PMID 21943617
- [Background] Dehghan M, Fatehi Poor A, Mehdipoor R, Ahmadinejad M. Does abdominal massage improve gastrointestinal functions of intensive care patients with an endotracheal tube?: A randomized clinical trial. Complement Ther Clin Pract. 2018 Feb;30:122-128. doi: 10.1016/j.ctcp.2017.12.018. Epub 2017 Dec 30. PMID 29389471
- [Background] McClurg D, Lowe-Strong A. Does abdominal massage relieve constipation? Nurs Times. 2011 Mar 29-Apr 4;107(12):20-2. PMID 21520798
- [Background] Arabul M, Kandemir A, Celik M, Alper E, Akpinar Z, Aslan F, Vatansever S, Unsal B. Impact of an information video before colonoscopy on patient satisfaction and anxiety. Turk J Gastroenterol. 2012;23(5):523-9. doi: 10.4318/tjg.2012.0416. PMID 23161296
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Ayan M, Tas U, Sogut E, Arici S, Karaman S, Esen M, Demirturk F. [Comparing efficiencies of diclofenac sodium and paracetamol in patients with primary dysmenorrhea pain by using Visual Analog Scale]. Agri. 2013;25(2):78-82. doi: 10.5505/agri.2013.42103. Turkish. PMID 23720082
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Kjeldsen HB, Klausen TW, Rosenberg J. Preferred Presentation of the Visual Analog Scale for Measurement of Postoperative Pain. Pain Pract. 2016 Nov;16(8):980-984. doi: 10.1111/papr.12344. Epub 2015 Aug 27. PMID 26310997
- [Background] Gagliese L, Weizblit N, Ellis W, Chan VWS. The measurement of postoperative pain: a comparison of intensity scales in younger and older surgical patients. Pain. 2005 Oct;117(3):412-420. doi: 10.1016/j.pain.2005.07.004. PMID 16153776
- [Background] Uysal N, Eser I, Akpinar H. The effect of abdominal massage on gastric residual volume: a randomized controlled trial. Gastroenterol Nurs. 2012 Mar-Apr;35(2):117-23. doi: 10.1097/SGA.0b013e31824c235a. PMID 22472671
- [Background] Altun Ugras G, Yuksel S, Isik MT, Tasdelen B, Dogan H, Mutluay O. Effect of abdominal massage on bowel evacuation in neurosurgical intensive care patients. Nurs Crit Care. 2022 Jul;27(4):558-566. doi: 10.1111/nicc.12575. Epub 2020 Nov 12. PMID 33179847
- [Background] Preece J. Introducing abdominal massage in palliative care for the relief of constipation. Complement Ther Nurs Midwifery. 2002 May;8(2):101-5. doi: 10.1054/ctnm.2002.0610. PMID 12188155
- Available data/document: Review — https://dergipark.org.tr/tr/download/article-file/117117
- Available data/document: Clinical Study Report — https://dergipark.org.tr/tr/download/article-file/29524